CLINICAL TRIAL: NCT05599633
Title: Effect of 12 Weeks Consumption of Sago Based Products in a Malaysian Diet on Glycaemic and Lipid Control in Diabetic Patients: a Double-Blind, Randomised, Parallel Controlled Trial
Brief Title: Effect of Sago-based Product on Glycaemic and Lipid Control in Diabetes
Acronym: SAGODM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sarawak General Hospital (Other)
Collaborators: CRAUN Research Sdn. Bhd. (Unknown)
Responsible Party: Principal Investigator, Xun Ting Tiong, Medical Officer, Sarawak General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CRC003-SAGODM
Record Dates: First submitted 2022-10-26; First posted 2022-10-31 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-04

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: diabetes mellitus; resistant starch; sago; Sarawak; glycemic control; lipid control
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Intervention (Sago starch) and control (corn starch) will be packed in individual aluminium sachets and will not be distinguishable from each other. The included subjects and investigators will be blinded from the study arm assignment. Randomisation and dispensation of the study starch will be done by the unblinded pharmacists only, who will not be involved in the care of the patients and study endpoint assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Arm (Experimental): Subjects who are randomised to Intervention Arm will be taking a drink containing 25g of Sarawak sago starch in 200mL of plain water. The subjects will take the drink twice daily i.e., within 30 minutes before lunch and dinner. On top of that, they will be counselled on diet recommendations for diabetes by a study dietitian at Visit 1 or baseline.
  Interventions: Dietary Supplement: Sago starch drink
- Control Arm (Placebo Comparator): Subjects who are randomised to Control Arm will be taking a drink containing 25g of corn starch in 200mL of water. The subjects will take the starch suspension twice daily i.e., within 30 minutes before lunch and dinner. On top of that, they will be counselled on diet recommendation for diabetes by a study dietitian at Visit 1 or baseline.
  Interventions: Dietary Supplement: Corn starch drink

INTERVENTIONS:
Dietary Supplement: Sago starch drink — Sarawak sago starch drink will be provided by CRAUN throughout the study. The starch drink will be supplied in sealed aluminium sachets. Each sachet contains 25g of study starch with cocoa flavouring.
  Arms: Intervention Arm
Dietary Supplement: Corn starch drink — Corn starch drink will be provided by CRAUN throughout the study. The starch drink will be supplied in sealed aluminium sachets. Each sachet contains 25g of study starch with cocoa flavouring.
  Arms: Control Arm

SUMMARY:
This will be a parallel, randomised, double-blind, controlled trial. Upon successful screening, subjects will be randomised to either intervention arm or control arm in a ratio of 1:1. The subjects will consume either a drink containing 25g of Sarawak sago starch (intervention) or 25g of corn starch (control) in approximately 200mL of water, two times a day, before lunch and dinner for 12 weeks, in addition to a standardised dietary counselling for diabetes given by the hospital dietitian at baseline. The study endpoints will be evaluated after 12 weeks of starch consumption.

DETAILED DESCRIPTION:
SAGODM trial is a parallel, randomised, double-blind, controlled trial on the effect of consuming sago starch for 12 weeks on glycaemic and lipid control in patients with type 2 diabetes mellitus. Diabetic patients who had HbA1C between 6.5% and 8.5% and had no change in the antidiabetic treatment for the past two months (primary inclusion criteria) were invited to participate in the trial. They were randomised to either the intervention arm or control arm in a ratio of 1:1. The subjects will consume either a drink containing 25g of Sarawak sago starch (intervention) or 25g of corn starch (control) in approximately 200mL of water, two times a day, before lunch and dinner for 12 weeks. They will receive standardised dietary counselling for diabetes given by the hospital dietitian at baseline. They will also be asked to record their dietary intake for three consecutive days every month. Blood samples will be taken at baseline and the last visit (post-12 weeks). The study endpoints will be evaluated after 12 weeks of starch consumption.

ELIGIBILITY:
Inclusion Criteria:

1. 18 - 70 years old
2. Individual diagnosed with type 2 diabetes for at least three months
3. Not on any antidiabetic medications or on lifestyle modification or taking a stable dose of oral hypoglycaemic agents, with no change of dose and regime for the past eight weeks
4. Has HbA1C values of 6.5 - 8.5% within 28 days before commencing the study
5. Able to complete the clinical study, and
6. Able to provide written informed consent

Exclusion Criteria:

1. History of allergy to sago starch or corn starch
2. History of allergy to any other ingredients in the study foods
3. Clinically significant, active and acute cardiovascular disease
4. Clinically significant, stage 4 - 5 (estimated glomerular filtration rate <30mL/min/1.73m2), chronic kidney failure
5. Clinically significant chronic liver disease or infection
6. Any malignancies
7. Regular use of hormone medications, anti-inflammatory medication, steroids, or other medications that might interfere with outcome measure
8. On a prescribed therapeutic diet
9. Taking part in weight loss programme
10. Clinically significant abnormal laboratory investigations
11. Other medical conditions or reasons, in the opinion of the Investigator or Research Physician, that make one unsuitable to join the study
12. Concurrent participation in other clinical studies involving intervention or treatment towards obesity, diabetes or impaired glucose
13. Pregnant or lactating mothers

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2024-01-19 (Actual); Study Completion 2024-01-20 (Actual)

PRIMARY OUTCOMES:
Change of HbA1C value | 12 weeks
  The change of HbA1C value at 12 weeks of intervention from baseline
Change of fasting blood glucose (FBG) level | 12 weeks
  The change of FBG level at 12 weeks of intervention from baseline
Change of homeostasis model assessment (HOMA) of insulin resistance (HOMA-IR) value | 12 weeks
  The change of HOMA of insulin resistant value at 12 weeks of intervention from baseline
Change of triglycerides level | 12 weeks
  The change of triglycerides level at 12 weeks of intervention from baseline
Change of total cholesterol level | 12 weeks
  The change of total cholesterol level at 12 weeks of intervention from baseline
Change of low density lipoprotein cholesterol (LDL-C) level | 12 weeks
  The change of LDL-C level at 12 weeks of intervention from baseline
Change of high density lipoprotein cholesterol (HDL-C) level | 12 weeks
  The change of HDL-C level at 12 weeks of intervention from baseline

SECONDARY OUTCOMES:
Change of inflammatory marker levels: high-sensitive c-reactive protein (hs-CRP) level | 12 weeks
  The change of hs-CRP level at 12 weeks of intervention from baseline
Change of inflammatory marker levels: interleukin 6 (IL-6) level | 12 weeks
  The change of IL-6 level at 12 weeks of intervention from baseline
Change of inflammatory marker levels: blood ferritin level | 12 weeks
  The change of blood ferritin level at 12 weeks of intervention from baseline
Change of total daily calorie intake | 12 weeks
  The change of total daily calorie intake at 12 weeks of intervention from baseline
Change of body weight/body mass index (BMI) | 12 weeks
  The change of BMI at 12 weeks of intervention from baseline
Change of body fat and visceral fat percentages | 12 weeks
  The change of body fat and visceral fat percentages at 12 weeks of intervention from baseline
Change of waist-hip ratio from baseline | 12 weeks
  The change of waist-hip ratio at 12 weeks of intervention from baseline
Change of blood pressure from baseline | 12 weeks
  The change of systolic and diastolic blood pressure at 12 weeks of intervention from baseline
Change of heart rate from baseline | 12 weeks
  The change of heart rate at 12 weeks of intervention from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Xun Ting Tiong, Principal Investigator — Clinical Research Centre Sarawak General Hospital
Locations (4):
- Malaysia (4):
  - Klinik Kesihatan Batu Kawah, Kuching, Sarawak
  - Klinik Kesihatan Jalan Masjid, Kuching, Sarawak
  - Klinik Kesihatan Tanah Puteh, Kuching, Sarawak
  - Sarawak General Hospital, Kuching, Sarawak

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] King TL, Bugam SH, Khoo SY, Tan SH, Yeo JJP, Tan SSN, Chan PY, Liew NK, Chunggat J, Tiong LL, Ibrahim AS, Tan FHS, Tiong XT. Effects of 12 Weeks consumption of sago starch on glycaemic and lipid control in patients with type 2 diabetes: A double-blind, randomised, parallel controlled trial. Clin Nutr ESPEN. 2025 Aug;68:300-308. doi: 10.1016/j.clnesp.2025.05.002. Epub 2025 May 8. PMID 40345654